CLINICAL TRIAL: NCT00687791
Title: Oculusgen (Ologen) Collagen Matrix Implant for Phaco-Trabeculectomy in Primary Glaucoma: A Case-Control Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pro Top & Mediking Company Limited (Industry)
Responsible Party: Assoc. Prof. Aung Tin, Singapore Eye Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mediking 0706
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Cataract; Glaucoma
Keywords: patients with cataract and glaucoma; ologen; oculusgen; collagen matrix; Phacotrabeculectomy; Aeon Astron; trabeculectomy; tissue engineering; mitomycin-C
MeSH Terms: conditions — Cataract; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 20 enrolled patients will be chosen according to the enrollment acceptance criteria. The evidence for the determination of enrolled patients shall be recorded, reviewed and approved. 2> Phacotrabeculectomy is performed.3> After completing phacotrabeculectomy, implant/place ologen™ Collagen Matrix on top of the scleral flap under the conjunctiva. For every inspection and observation, the detailed description and/or inspection data shall be recorded. If any unwanted adverse event is observed during inspection and observation, it shall be recorded and be reported to the investigation conductor.
  Interventions: Device: ologen™ Collagen Matrix Implant as an aid in phacotrabeculectomy surgery

INTERVENTIONS:
Device: ologen™ Collagen Matrix Implant as an aid in phacotrabeculectomy surgery — Study of the safety and effectiveness of the ologen™ Collagen Matrix Implant as an aid in phacotrabeculectomy surgery
  Other Names: OculusGen (ologen™)

SUMMARY:
The objective of this study is to determine the safety and effectiveness of the OculusGen™ (ologen) Biodegradable Collagen Matrix Implant in hacotrabeculectomy surgery. The primary endpoint is to prove the effectiveness via the reduction of IOP, and the secondary endpoint is to prove the safety via the incidence of complications and adverse events.

DETAILED DESCRIPTION:
Ologen™ Collagen Matrix is indicated for creating a mature bleb structure to facilitate aqueous outflow for the reduction of elevated intraocular pressure in patients with glaucoma, following traditional filtering surgery (trabeculectomy)

Within 60 days from the time of implantation, ologen™ Collagen Matrix is totally degraded. Postoperatively, mild inflammation may be seen and anti- inflammatory agents are prescribed

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over.
2. At least one eye diagnosed with glaucoma and receiving maximally tolerated medical therapy.
3. Visually significant cataract with visual acuity of less than or equal to 6/12.
4. Subject able and willing to cooperate with investigation plan.
5. Subject willing to sign informed consent form.

Exclusion Criteria:

1. Known allergic reaction to collagen.
2. Subject is on Warfarin and discontinuation is not recommended.
3. Subject with normal tension glaucoma or aphakic glaucoma.
4. Subject with corneal disease.
5. Participation in an investigational study during the 30 days proceeding phacotrabeculectomy.
6. Ocular infection within 14 days prior to phacotrabeculectomy.
7. Pregnant or breast-feeding women.
8. Monocular subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to prove the effectiveness via the reduction of IOP. | 180 days

SECONDARY OUTCOMES:
the secondary endpoint is to prove the safety via the reduction of complications. | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Aung Tin, PhD MD, Study Chair — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore